CLINICAL TRIAL: NCT02364687
Title: Optimisation and Quantification of Contrast Enhanced Computed Tomography
Brief Title: Optimisation and Quantification of Contrast Enhanced Computed Tomography Myocardial Fibrosis Imaging
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 13/SS/0152
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2023-06-27 (Actual); Status verified 2022-06

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: Participants will have previously had an MRI scan and will undergo a CT scan.
  Interventions: Radiation: Computed tomography late enhancement imaging

INTERVENTIONS:
Radiation: Computed tomography late enhancement imaging

SUMMARY:
Detecting scarred heart muscle is important to diagnose and treat of a wide variety of heart conditions. Magnetic resonance imaging (MRI) can assess scarred heart muscle but it is time consuming, contraindicated for some patients and not tolerated by others. Computed tomography (CT) imaging has the potential to provide a rapid comprehensive assessment of the heart. This study will assess CT imaging of the heart muscle of patients who have previously undergone MRI of their heart. Using a state of the art CT scanner the investigators will develop a low radiation dose protocol to identify scarred heart muscle. The investigators will use and develop software techniques to analyse these images. This will enable us to develop a new way to identify and measure scarred heart muscle that will benefit patients with heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Presence of late enhancement on magnetic resonance imaging

Exclusion Criteria:

* age less than 40
* inability or unwillingness to undergo CT
* renal failure (serum creatinine >200 umol/l or estimated glomerular filtration rate <30 ml/min)
* hepatic failure
* allergy to iodinated contrast
* pregnancy
* breast feeding
* inability to undergo informed consent
* fast atrial fibrillation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have previously undergone magnetic resonance imaging which showed myocardial late enhancement.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Myocardial late enhancement | Immediate
  The amount of myocardial late enhancement measured on computed tomography as compared to magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Williams, Principal Investigator — University of Edinburgh, NHS Lothian